CLINICAL TRIAL: NCT06848426
Title: A Clinical Study of Xingbaiji Formula in Combination with Chemotherapy and Sintilimab As First-Line Treatment for Metastatic Multi-Target Mutation-Negative Non-Small Cell Lung Cancer
Brief Title: Xingbai Ji Formula Combined with Chemotherapy and Sintilimab in Metastatic Multi-Target Mutation-Negative Non-Small Cell Lung Cancer: a Clinical Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jiangxi Provincial People's Hopital (Other)
Responsible Party: Principal Investigator, Weirong Yao, Chief Physician, Jiangxi Provincial People's Hopital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202510200
Record Dates: First submitted 2025-02-18; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2024-12

CONDITIONS: Non-Small Cell Lung Cancer; Non-small Cell Lung Cancer Recurrent; Non-small Cell Lung Cancer Stage IIIB; Non-small Cell Lung Cancer Stage IV; Non-small Cell Lung Cancer Metastatic
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Arm (No Intervention)
- Intervention Arm (Experimental)
  Interventions: Drug: Xingbaiji Formula

INTERVENTIONS:
Drug: Xingbaiji Formula — Patients were randomized into two groups:
  Control Group:
  Non-squamous NSCLC: Sintilimab (200 mg) combined with pemetrexed + cisplatin/carboplatin, administered intravenously (IV) every 3 weeks (Q3W) for 4 cycles. After 4 cycles, maintenance therapy with sintilimab (200 mg Q3W, up to 24 months) + pemetrexed Q3W continued until disease progression, intolerable toxicity, death, or voluntary withdrawal.
  Squamous NSCLC: Sintilimab (200 mg) combined with gemcitabine + cisplatin/carboplatin, IV Q3W for 4-6 cycles. Post-induction, sintilimab (200 mg Q3W) maintenance continued until progression, intolerance, or ≤2 years of treatment.
  Experimental Group:
  The control regimen plus Xingbaiji Formula:
  Xingbaiji Granule 1: 10 g/bag, dissolved in warm water, 1 bag twice daily (morning and evening) after meals.
  Xingbaiji Granule 2: 5 g/bag, dissolved in warm water, 1 bag twice daily (morning and evening) after meals.
  Arms: Intervention Arm

SUMMARY:
Clinical Trial Protocol

Primary Objective:

To evaluate the efficacy of the Xingbaiji Formula combined with chemotherapy and Sintilimab as first-line therapy in patients with recurrent or metastatic Stage IIIB-IV EGFR/ALK/ROS-1 mutation-negative non-small cell lung cancer (NSCLC), using Objective Response Rate (ORR) of tumor lesions as the primary endpoint.

Secondary Objectives:

To assess secondary endpoints including Progression-Free Survival (PFS), Quality of Life (QoL), immune-related indicators, and safety profile (e.g., incidence of adverse events), and to further evaluate the efficacy and safety of the combination therapy.

Randomized Group Allocation:

Participants will be randomly assigned to two groups:

Control Group

Regimen for Advanced Non-Squamous NSCLC:

Drugs and Dosage:

Sintilimab 200mg + Pemetrexed + Cisplatin/Carboplatin via intravenous infusion, administered every 3 weeks (Q3W) for 4 cycles.

After completion of 4 cycles, patients enter the maintenance phase: Sintilimab 200mg Q3W (up to 24 months) + Pemetrexed Q3W until disease progression, intolerable toxicity, death, or voluntary withdrawal.

Regimen for Advanced Squamous NSCLC:

Drugs and Dosage:

Sintilimab 200mg + Gemcitabine + Cisplatin/Carboplatin via intravenous infusion, Q3W for 4-6 cycles.

Post-treatment, patients receive Sintilimab 200mg Q3W maintenance until disease progression, intolerability, or completion of 2 years of Sintilimab therapy.

Experimental Group Control Group Regimen + Xingbaiji Formula

Xingbaiji Formula Dosage:

1. Granule No. 1: 10g/bag, dissolved in warm water. Administration: 1 bag orally, twice daily (morning and evening), after meals.
2. Granule No. 2: 5g/bag, dissolved in warm water. Administration: 1 bag orally, twice daily (morning and evening), after meals. Treatment Duration: Both granules are taken concurrently with chemotherapy for 6 months, then discontinued.

DETAILED DESCRIPTION:
Randomized Clinical Trial on Xingbaiji Formula Combined with Chemotherapy and Sintilimab as First-Line Treatment for Recurrent/Metastatic Stage IIIB-IV EGFR/ALK/ROS-1 Mutation-Negative Non-Small Cell Lung Cancer Primary Objective: To evaluate efficacy by measuring Objective Response Rate (ORR) in patients receiving Xingbaiji Formula combined with chemotherapy and Sintilimab.

Secondary Objectives: To assess Progression-Free Survival (PFS), Quality of Life (QoL), immune-related biomarkers, safety, and adverse event rates.

Study Arms Control Group

Non-squamous NSCLC:

Sintilimab 200mg + Pemetrexed + Cisplatin/Carboplatin (IV, Q3W for 4 cycles). After induction, maintenance with Sintilimab 200mg Q3W (≤24 months) + Pemetrexed Q3W until disease progression, toxicity, or withdrawal.

Squamous NSCLC:

Sintilimab 200mg + Gemcitabine + Cisplatin/Carboplatin (IV, Q3W for 4-6 cycles). Maintenance with Sintilimab 200mg Q3W until progression or maximum 2 years.

Experimental Group

Control Regimen + Xingbaiji Formula:

Xingbaiji Granule 1 (10g/sachet): Dissolved in warm water, 1 sachet twice daily (morning/evening, post-meal).

Xingbaiji Granule 2 (5g/sachet): Dissolved in warm water, 1 sachet twice daily (morning/evening, post-meal).

Duration: Concurrent with chemotherapy for 6 months, then discontinued.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent.
2. Age: 18-75 years, regardless of gender.
3. Histologically or cytologically confirmed non-small cell lung cancer (NSCCC), including adenocarcinoma, squamous cell carcinoma, or large cell carcinoma, with negative EGFR, ALK, and ROS-1 mutations confirmed by next-generation sequencing (NGS). Stage IIIB-IV NSCLC as per AJCC 8th edition staging criteria (required evaluations: neck contrast-enhanced CT or ultrasound, chest contrast-enhanced CT, abdominal contrast-enhanced CT or ultrasound, brain contrast-enhanced MRI, bone scan, or whole-body PET/CT).
4. ECOG performance status ≤2 and life expectancy ≥3 months.
5. Histologically or cytologically documented ineligibility for EGFR, ALK, or ROS-1 targeted therapies (written evidence required).
6. At least one measurable lesion per RECIST v1.1. Lesions within prior radiation fields or post-local treatment may be selected if progression is confirmed.
7. No prior systemic anti-tumor therapy for advanced disease. Adjuvant chemotherapy is permitted if ≥6 months have elapsed between recurrence and the last dose.

Exclusion Criteria:

1. History of or concurrent other malignancies (excluding non-invasive tumors such as cured basal cell carcinoma of the skin, cervical carcinoma in situ, etc.);
2. Individuals with allergic reactions to the Xingbaiji formula;
3. Patients with mixed small cell lung cancer or those with a small cell lung cancer component;
4. Severe mental illness or cognitive impairment that would impede compliance with study protocols or follow-up requirements;
5. Pregnant or lactating women (a pregnancy test must be performed to exclude pregnancy; women of childbearing age must agree to use effective contraception during the study);
6. Presence of any major illness or significant laboratory abnormalities that may interfere with receiving Xingbaiji formula, chemotherapy, or immunotherapy; 7Any other conditions deemed by the investigators to render participation in the trial inappropriate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03-10 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | six months

SECONDARY OUTCOMES:
Progression-Free Survival(PFS) | 1 year
Disease Control Rate（DCR） | six months

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangxi Provincial People's Hospital, Nanchang, Jiangxi, China